CLINICAL TRIAL: NCT02925884
Title: The Effect of Computer Eyewear on Viewing Comfort and Performance in Office Work
Brief Title: Effects of Gunnar Computer Glasses on Viewing Comfort and Performance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor failed to provide financial support as promised.
Sponsor: Pacific University (Other)
Collaborators: Gunnar Optiks (Other)
Responsible Party: Principal Investigator, Yu-Chi Tai, Research Scientist, Pacific University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PUIRB075-13; Gunnar2013 (Other Grant/Funding Number: Gunnar Optiks)
Record Dates: First submitted 2013-06-17; First posted 2016-10-06 (Estimated); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye; Eye Strain; Visual Acuity; Color Perception
Keywords: Computer Glasses; Dry eye; Eye strain; Gunnar Glasses
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimenter: Gunnar OTC Glasses, Then Control (Experimental): On Visit 1, after the screening and baseline measurements, participants were given a pair of Gunnar OTC glasses (Intervention 1) and asked to work on the computer with the glasses for at least 4 hours for 5+/-2 days of adaptation (Habituation 1).
  On Visit 2, they performed the designated computer tasks with the glasses to complete the Gunnar condition. Then they were asked to work on the computers for at least 4 hours without any glasses (Intervention 2) for another 5+/-2 days (Habituation 2).
  On Visit 3, they performed the same tasks without any glasses to complete the Control condition. Then Participants responded if they prefer wearing the Gunnar OTC Glasses when working on a computer.
  Interventions: Device: Gunnar OTC Glasses
- Experimenter: Control, Then Gunnar OTC Glasses (Experimental): On Visit 1, after the screening and baseline measurements, participants were told to work on the computer for at least 4 hours without glasses (Intervention 1) for 5+/-2 days of adaptation (Habituation 1).
  On Visit 2, they performed the designated computer tasks without glasses to complete the Control condition. Then they were given a pair of Gunnar OTC Glasses to wear (Intervention 2) while working on the computers for 4+ hours daily for another 5+/-2 days (Habituation 2).
  On Visit 3, they performed the same tasks with the Gunnar glasses to complete the Gunnar condition. Then Participants responded if they prefer wearing the Gunnar OTC Glasses when working on a computer.
  Interventions: Device: Gunnar OTC Glasses

INTERVENTIONS:
Device: Gunnar OTC Glasses — Gunnar Over-the-Counter Computer Glasses have optical power of 0.5 diopters for reducing accommodation demands at a typical computer-viewing distance. The lens also have a partially transmissive yellow tinting and anti-reflective coating for filtering part of the spectral peaks in typical fluorescent or incandescent light. The frame has a wrape-around design meant to reduce air flow in the vicinity of the eyes.

SUMMARY:
The proposed study aims to test if Gunnar computer glasses provide any advantages, in comparison to no glasses, on the following aspects in computer-related office work:

* Any enhancement on the visual performance of the basic visual function, including visual acuity, contrast sensitivity, color discrimination, etc.
* Any enhancement on the visual performance of typical office work, including reading, word-spelling check, number searching, or target identification.
* Any benefit in objective viewing comfort measured with viewing distance, blink frequency, post-viewing pupil size.
* Any benefit in subjective viewing comfort reflected on the questionnaire of viewing symptom survey.
* Any benefit in viewing comfort and visual performance with increased environmental ventilation or under the strong glare.
* Any benefit in life quality from daily wearing (e.g., better comfort or sleep quality).

DETAILED DESCRIPTION:
<Introduction>

When performing near work, one must focus at (accommodate) and point toward (converge) at a closer distance and constantly re-focus the eyes to see small text and images with clarity. Sustaining such efforts can lead to eye fatigue and eye strain, among a host of vision problems. Most visual tasks on a screen also demand heightened visual concentration, and this decreases blink rate. Working in a heated or air-conditioned office environment leads to over-evaporation of the tear film, and lipid deficiency, irritation, and dryness to the corneal surface are expected. Disruptive glare from excessive screen reflection and ambient lighting also deteriorates the image quality and heaps on viewing discomfort. Extensive screen viewing also exacerbates discomfort in people with existing vision problems like eye muscle imbalance, astigmatism, farsightedness, and presbyopia. Since technology is almost unavoidable to modern life, preventions should be taken to lessen the total toll on the eyes and visual system. Gunnar computer glasses address the above issues by providing mild yellow tint anti-reflection coating to shield the harmful blue light and lessen strong glare. The glasses also have a small amount of magnification (+0.5 D) to enhance acuity. The curved frame is designed to retain moisture and reduce dry eye symptoms. All these special characters are devised to enhance visual performance and minimize eye fatigue and visual discomfort in digital viewing. The current study aimed to validate the benefits mentioned above.

Gunnar over-the-counter (OTC) computer glasses adopt yellow lenses to cut off the active short wavelength and lessen the bright glare, which often induces the detrimental effect caused by excessive illumination or intense scattered reflection. While the benefit of glare reduction is well received, the benefit on visual performance has been inconclusive. Some studies reported a significant enhancement in contrast sensitivity, but some failed to see any improvement in visual acuity and contrast sensitivity, even with color distortion. Without argument, tinted lenses reduce the transmittance of the visible spectrum and change the visible color to a certain degree. However, there has been a report that reducing the retinal illumination level does not necessarily lead to reduced brightness; instead, the visual system automatically adjusts for the illumination discounting, possibly with the help of increased pupil size. In addition, with the decrement of blue lights arriving at the eyes, both scattered reflection and chromatic aberration are reduced. Together, it is reasonable to believe that the visual acuity, contrast sensitivity, and chromatic discrimination will not suffer and may, instead, benefit from the filter of yellow lenses. These basic visual functions may, in turn, lead to enhancement in general visual performance such as routine office work. These will be tested in the proposed study.

The current study tested if Gunnar's OTC computer glasses provide any advantages, in comparison to no glasses, on the following aspects in computer-related office work:

* Any enhancement on the visual performance of the basic visual function, including visual acuity, contrast sensitivity, color discrimination, etc.
* Any enhancement on the visual performance of typical office work, including reading, word-spelling check, number searching, or target identification.
* Any benefit in preventing dry eye by measuring the humidity outside and inside the frame (only in the visit with Gunnar glasses) and the tear film break-up time after viewing for a prolonged period.
* Any benefit in objective viewing comfort measured with viewing distance, blink frequency, post-viewing pupil size.
* Any benefit in subjective viewing comfort reflected on the questionnaire of viewing symptom survey.
* Any benefit in viewing comfort and visual performance with increased environmental ventilation.
* Any benefit in viewing comfort and visual performance with increased environment under the intense glare.
* Any benefit in life quality from daily wearing (e.g., viewing comfort, sleep quality, or quantity due to the amount of stimulation from blue light)?
* Their willingness to purchase (select) the tested Gunnar OTC glasses and the price willing to pay for.

<Study design>

Thirty-four subjects, age 18 to 42, were planned to be recruited. This sample size is based on a priori power analysis with 80% and a medium effect size at alpha equal to 0.05. Subjects will be stratified into four age groups. An about equal number (8±1) of subjects should have been recruited for each group:

* 18-23 yr old
* 24-29 yr old
* 30-35 yr old
* 36-42 yr old

Each subject was scheduled for three visits: Visit 1 for screening and consenting, visit 2 for lab test after treatment 1, and visit 3 for lab test after treatment 2. Between visits was an adaptation period for the assigned treatment.

Visit 1: A screening visit

* Day 1, when a subject first joins the study
* Obtain informed consent and screening measurements (VA, contrast sensitivity, tear film break-up time as dry eye measurement, Dry eye questionnaire (OSDI), viewing symptom survey (VSS), history of dry eye, and computer work behavior).
* At the end of the visit, half of the subjects were given a pair of Gunnar OTC glasses for adaptation for 3 - 7 days; the other half were given no treatment. All subjects were told to work in front of a computer for at least 4 hours a day, with the assigned glasses if given.

Adaptation 1:

- Starting on Day 1, for 3 to 7 days, the subject was asked to work in front of computers for at least 4 hours each day with assigned treatment 1.

Visit 2: Lab test for treatment 1

* On a day between day four and day 8 convenient to the subject, the subject came to the lab with the assigned glasses condition.
* Baseline measurements will be taken, followed by a few visual tasks under three viewing conditions. The subject was asked to fill out the VSS, given a break, before being tested on another round of tasks under a different viewing condition.
* The total testing time is about 70 minutes for each condition and about 4 hours to complete the visit.
* The lab testing procedure is described below.
* At the end of visit 2, treatment was alternated for another 3-7 days of adaptation.

Adaptation 2 with treatment 2:

- Starting on the day of Visit 2 after the test, the subject adapts to the second treatment (with Gunnar glasses or without any glasses) for another 3 to 7 days.

Visit 3: Lab test for treatment 2

* The same procedure of Visit 2 was repeated.
* Subject was asked to rate their preference of wearing the Gunnar Glasses over no-glasses when performing computer tasks.
* After this visit, the study was completed for the subject.

Details of lab testing procedures:

* The study adopted a crossover design. Each subject went through three viewing conditions (control, bright light, strong ventilating) based on a Latin Square order.

  1. In the control condition, the subject will perform all tasks under regular office lighting (500 lux) and the default lab ventilation condition.
  2. In the bright light condition, the ambient light will be increased to 1500 lux.
  3. In the strong ventilation condition, a ceiling fan will be positioned on top of the subject at the ceiling light location to increase the airflow.

     Visual performance tasks:
* Baseline measurements (10 min): Upon arrival, the subject was asked to fill out VSS and OSDI. Measurements of dry eye condition, pupil size, accommodation status, and blink rate were taken as the baseline for a visit.
* Under viewing condition 1:

  1. Visual tasks (60 minutes): Visual acuity, contrast sensitivity, color perception, visual search of numbers among a number matrix, low-contrast target search, text reading, and spelling check were performed by a fixed order.
  2. Post-task measurements of dry eye measure (Tear break uptime), pupil size, accommodation, and blink rate, as well as VSS were taken.
* Break time of 5-10 minutes.
* Repeat the above procedures for the other two viewing conditions.
* Total time for one lab visit was about 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 18 to 42 years old.
* Subjects must have a normal color vision (be able to identify the numbers in the color blind test.
* Subjects' near and far visual acuity with the better eye needs to be 20/25 or better (measured with a vision chart). Subjects can wear contact lenses (but not glasses) if usually wear them while working on computers.
* Subjects must routinely work on a computer or digital display for an average of 4 hours or more each day.
* Subjects can communicate in English fluently and are used to read English documents on a computer.
* Subjects must have a valid tax number or social security number to receive monetary compensation.

Exclusion Criteria:

* The difference in the prescription for both eyes is equal to or larger than 2 Diopters.
* Subjects have a cataract or have had cataract surgery.
* Subjects are sensitive to lights (photosensitivity).
* Subjects have prior incidents or are known to have claustrophobia.
* Subjects have been diagnosed with oculomotor diseases or central nervous system diseases, or with developmental, neurological, or psychiatric disorders (e.g., attention deficit hyperactivity disorder, autism, mental retardation).

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chi Tai, PhD, Principal Investigator — Pacific University
Locations (1):
- Vision Performance Institute, 129 Scott Hall, Pacific University, Forest Grove, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- See also: Summary of the current findings — https://pacificu.box.com/s/3l9xdwrrohp1i48ul0frbxdo5m6uhg3m

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 participants were screened and enrolled between June 28, 2013 and September 30th, 2013 in the Vision Performance Institute research lab in Scott Hall 129 at Pacific University Forest Grove Campus.
Pre-assignment Details: (not apply)
Groups:
- Gunnar OTC Glasses, Then Control: On Visit 1, participants were screened to meet the recruitment criteria, and their baseline ocular conditions were measured. At the end of the visit, they were given Intervention 1 of a pair of Gunnar OTC glasses to wear while working on computers for 4+ hours each day for the following 5+/-2 days (Habituation 1). On Visit 2, their visual performance and ocular conditions were measured with the Gunnar glasses. Then they were told to work on the computer without any glasses (Intervention 2) for 4+ hours each day for another 5+/-2 days (Habituation 2). On Visit 3, they return to the lab for the same tests without glasses.
- Control, Then Gunnar OTC Glasses: At Visit 1, participants were screened to meet the recruitment criteria, and their baseline ocular conditions were measured. At the end of the visit, they were told to work on computers WITHOUT any glasses (Intervention 1) for 4+ hours each day for the following 5+/-2 days of Habituation 1. On Visit 2, their visual performance and ocular conditions were measured WITHOUT any glasses. Then they were given Intervention 2 of a pair of the Gunnar OTC glasses and asked to wear it while working on the computer for 4+ hours per day for another 5+/-2 days (Hibuation 2). On Visit 3, they return to the lab for the same tests with Gunnar OTC glasses on.
Period: Visit 1: Screening & Give Intervention 1
Arm/Group | Gunnar OTC Glasses, Then Control | Control, Then Gunnar OTC Glasses
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0
Period: Habituation 1
Arm/Group | Gunnar OTC Glasses, Then Control | Control, Then Gunnar OTC Glasses
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0
Period: Visit 2: Lab Test & Give Intervention 2
Arm/Group | Gunnar OTC Glasses, Then Control | Control, Then Gunnar OTC Glasses
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0
Period: Habituation 2
Arm/Group | Gunnar OTC Glasses, Then Control | Control, Then Gunnar OTC Glasses
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0
Period: Visit 3: Lab Test 2
Arm/Group | Gunnar OTC Glasses, Then Control | Control, Then Gunnar OTC Glasses
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control, Then Gunnar OTC Glasses: On Visit 1, participants were screened to meet the recruitment criteria, and their baseline ocular conditions were measured. At the end of the visit, they were told to work on the computer for at least 4 hours without glasses (Intervention 1) for 5+/-2 days of adaptation (Habituation 1). On Visit 2, their visual performance and ocular conditions were measured without glasses to complete the Control condition. Then they were given a pair of Gunnar OTC Glasses to wear (Intervention 2) while working on the computers for 4+ hours daily for another 5+/-2 days (Habituation 2). On Visit 3, they performed the same tasks with the Gunnar glasses to complete the Gunnar condition.
- Total: Total of all reporting groups
Arm/Group | Gunnar OTC Glasses, Then Control | Control, Then Gunnar OTC Glasses | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 9 | 12 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Rating of Gunnar Computer Glasses Preference
Description: At the end of the study in Visit 3, subjects were asked to respond if they felt the Gunnar TC Glasses improved their computer viewing comfort and visual performance (choose between "Yes" and "No").
Time Frame: at the end of the study in Visit 3, up to day 16
Population: All participants receiving both intervention were measured and included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Age Group 1 (18-23 yo): At the end of the study (Visit 3), participants of the youngest age group (18-23 year-olds) were asked to respond if they felt the Gunnar TC Glasses improved their computer viewing comfort and visual performance (choose between "Yes" and "No"). They received the Gunnar OTC Glasses either as Intervention 1 or Intervention 2 to wear during the Habituation period and the immediate following lab testing time.
- Age Group 2 (24-29 yo): At the end of the study (Visit 3), participants of the second age group (24-29 year-olds) were asked to respond if they felt the Gunnar TC Glasses improved their computer viewing comfort and visual performance (choose between "Yes" and "No"). They received the Gunnar OTC Glasses either as Intervention 1 or Intervention 2 to wear during the Habituation period and the immediate following lab testing time.
- Age Grup 3 (30-35 yo): At the end of the study (Visit 3), participants of the third age group (30-35 year-olds) were asked to respond if they felt the Gunnar TC Glasses improved their computer viewing comfort and visual performance (choose between "Yes" and "No"). They received the Gunnar OTC Glasses either as Intervention 1 or Intervention 2 to wear during the Habituation period and the immediate following lab testing time.
- Age Group 4 (36-42 yo): At the end of the study (Visit 3), participants of the fourth (and the oldest) age group (36-42 year-olds) were asked to respond if they felt the Gunnar TC Glasses improved their computer viewing comfort and visual performance (choose between "Yes" and "No"). They received the Gunnar OTC Glasses either as Intervention 1 or Intervention 2 to wear during the Habituation period and the immediate following lab testing time.
Arm/Group | Age Group 1 (18-23 yo) | Age Group 2 (24-29 yo) | Age Grup 3 (30-35 yo) | Age Group 4 (36-42 yo)
Number analyzed (Participants) | 9 | 9 | 8 | 9
Participants
  Participant response : Yes | 6 | 7 | 8 | 9
  Participant response : No | 3 | 2 | 0 | 0

2. Secondary Outcome: Subjective Viewing Discomfort Rating
Description: Subjective rating of viewing comfort on the Viewing Symptom Survey (15 items, 5-pt Likert scale, 0: no discomfort; 4: extremely discomfort). Factor Analysis reduced the information dimension from 15 items to 5 factors:
  1. Decreased cognitive function: sleepy, can't concentrate, can't think clearly, difficulty to remember
  2. Eyestrain: eye strain, tired eyes
  3. Physical discomfort: body discomfort, neckache, headache
  4. Decreased visual function: blurry, double vision, can't focus, moving text
  5. Poor balance: vertigo, dizzy A factor score is a linear transformation of the variables with weights. Its unit is arbitrary and meaningless; no min or max. However, as the values (correlation between variable and factor) in the Structure Matrix are positive, the sign of the factor is the same as the variables. Positive larger values mean more discomfort. A linear mixed model compares the relative impact of the interventions (Gunnar OTC glasses vs. Control_No glasses) on each factor.
Time Frame: Data were collected at the end of Visit 2 (at least 3 days after Visit 1, between Day 4 and Day 8) and Visit 3 (at least 3 days after Visit 2, up to Day 16).
Population: All participants who received at least one Intervention were included in the analysis.
Measure: Mean (Standard Error); unit: factor score
Groups:
- Gunnar OTC Glasses: Participants who received the Gunnar OTC Glasses (either as Intervention 1 or Intervention 2) to wear both during the Habituation period (either Habituation 1 or Habituation 2) and the following lab testing time (either Visit two or Visit 3).
- Control: Participants who received NO Glasses (either as Intervention 1 or Intervention 2) to wear both during the Habituation period (either Habituation 1 or Habituation 2) and the following lab testing time (either Visit 2 or Visit 3).
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
factor score
  Decreased cognitive function | -0.128 (0.109) | 0.154 (0.111)
  Eyestrain | -0.228 (0.099) | 0.239 (0.101)
  Physical discomfort | 0.132 (0.114) | -0.117 (0.115)
  Decreased visual function | -0.187 (0.115) | 0.197 (0.117)
  Poor balance | -0.107 (0.112) | 0.109 (0.113)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Null hypothesis: No difference between the Gunnar OTC Condition and the Control Condition on the factor score of Decreased Cognitive Functions; Test type: Superiority; p = 0.011, Mixed Models Analysis
Statistical Analysis 2: Comparison: Gunnar OTC Glasses vs Control; Null hypothesis: No difference between the Gunnar OTC Condition and the Control Condition on the factor score of Eyestrain; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Gunnar OTC Glasses vs Control; Null hypothesis: No difference between the Gunnar OTC Condition and the Control Condition on the factor score of Physical Discomfort; Test type: Superiority; p = 0.009, Mixed Models Analysis
Statistical Analysis 4: Comparison: Gunnar OTC Glasses vs Control; Null hypothesis: No difference between the Gunnar OTC Condition and the Control Condition on the factor score of Deceased Visual Function; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 5: Comparison: Gunnar OTC Glasses vs Control; Null hypothesis: No difference between the Gunnar OTC Condition and the Control Condition on the factor score of Poor Balance; Test type: Superiority; p = 0.28, Mixed Models Analysis

3. Secondary Outcome: Visual Acuity
Description: The participant's ability to identify high-contrast objects was measured in Visits 2 and 3. Measurements were recorded in the logarithmic Measure of Angle of Resolution (logMAR) scale, in which each 'line' of the symbols on a vision chart corresponds to a unit of 0.1 and represents a 10-fold difference in acuity compared to the adjacent line of the vision. Normal (6/6 or 20/20) vision in Snellen notation equals 0.0 logMAR (logarithmic of 1.0 arc minute or 1/60 of a degree). A negative logMAR value means better than normal (20/20) vision, and a smaller logMAR represents better vision in distinguishing finer details.
Time Frame: during Visit 2 (at least 3 days after Visit 1, between Day 4 and Day 8) and Visit 3 (at least 3 days after Visit 2, up to Day 16)
Population: All participants received at least one Intervention were included in the analysis.
Measure: Mean (Standard Error); unit: logMAR
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
logMAR | -0.474 (0.002) | -.0474 (0.002)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Test type: Superiority; p = 0.903, Mixed Models Analysis

4. Secondary Outcome: Color Perception
Description: Participants' best performance in discriminating the number of color saturation levels was measured during visits 2 and 3. In each trial, six circles of the same color in 1-6 shades were presented. Participants responded with the number of color shades presented. Four colors (red, green, blue, and gray) were tested and analyzed separately. Performance in gray was used as the covariate for analysis.
Time Frame: during Visit 2 (at leadays after Visit 1, between Day 4 and Day 8) and Visit 3 (at least 3 days after Visit 2, up to Day 16)
Population: All participants received both interventions were included in the analysis.
Measure: Mean (Standard Error); unit: color saturation shades
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
color saturation shades
  Red | 2.952 (0.059) | 3.102 (0.059)
  Green | 2.935 (0.046) | 2.887 (0.045)
  Blue | 3.404 (0.075) | 3.399 (0.075)
  Gray | 5.320 (0.961) | 5.000 (0.962)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Null hypothesis: No difference between the Gunna OTC Glasses condition and the Control condition on Red Color Perception; Test type: Superiority; p = 0.009, Mixed Models Analysis
Statistical Analysis 2: Comparison: Gunnar OTC Glasses vs Control; Null hypothesis: No difference between the Gunna OTC Glasses condition and the Control condition on Green Color Perception; Test type: Superiority; p = 0.446, Mixed Models Analysis
Statistical Analysis 3: Comparison: Gunnar OTC Glasses vs Control; Null hypothesis: No difference between the Gunna OTC Glasses condition and the Control condition on Blue Color Perception; Test type: Superiority; p = 0.953, Mixed Models Analysis

5. Secondary Outcome: Spelling Check Accuracy
Description: subject's accuracy in spelling check.
Time Frame: Performance was measured during visit 2 (at least 3 days after Visit 1, between Day 4 and Day 8) and visit 3 (at least 3 days after Visit 2, up to Day 16).
Population: All participants received bth inventions were included in the analysis.
Measure: Mean (Standard Error); unit: percentage of accuracy
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
percentage of accuracy | .778 (.029) | .812 (.029)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Test type: Superiority; p = 0.266, Mixed Models Analysis

6. Secondary Outcome: Dry Eye Measurements (1): Tear Film Break-up Time (Seconds)
Description: Tear film break-up time (TBUT) measures the duration the tear covers the cornea surface fully until it evaporates. It reflects the stability of the tear film and is commonly used in clinics to check for evaporative dry eye syndrome. In testing for TBUT, sodium fluorescein dye is added to the eye, and the tear film is observed under the slit lamp while the patient avoids blinking until tiny dry spots develop. Larger numbers mean the tear stays on the cornea surface longer and is less severe for dry eye symptoms. Usually, TBUT values range from 3-132 seconds (average 27 seconds). TBUT less than 10 seconds suggests an abnormal tear film, 5-10 seconds considered marginal, and less than 5 seconds indicative of dry eye.
Time Frame: during Visit 2 (at least 3 days after Visit 1, between Day 4 and Day 8) and Visit 3 (at least 3 days after Visit 2, upto Day 16)
Population: All participants receiving both interventions were included in the analysis.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
seconds | 6.018 (0.347) | 6.438 (0.336)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Test type: Superiority; p = 0.424, Mixed Models Analysis

7. Secondary Outcome: Contrast Sensitivity
Description: The participant's ability to identify low-contrast objects was measured in Visits 2 and 3.
  A letter contrast sensitivity test by M&S Technology measures the subject's ability to detect objects without a clear outline and distinguish them from their background. The M&S Letter Contrast Sensitivity Test uses standard Snellen and Sloan Letters presented at contrast levels from 100% to 0.8%, with smaller numbers indicating better performance (better contrast sensitivity).
Time Frame: as for outcome 3
Population: All participants received at least one Intervention were included in the analysis.
Measure: Mean (Standard Error); unit: contrast ratio expressed in "%"
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
contrast ratio expressed in "%" | 1.115 (0.024) | 1.145 (0.024)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Test type: Superiority; p = 0.343, Mixed Models Analysis

8. Secondary Outcome: Spelling Check Speed (Words Per Minute, WPM)
Description: This measures the subject's speed (words per minute) in spelling check. Higher values mean better performance or more words being checked within one minute.
Time Frame: as for outcome 5
Population: All participants received bth inventions were included in the analysis.
Measure: Mean (Standard Error); unit: words per minute
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
words per minute | 178.892 (7.427) | 183.319 (7.285)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Test type: Superiority; p = 0.489, Mixed Models Analysis

9. Secondary Outcome: Dry Eye Measurements 2: Tear Osmolarity Index Measured With TearLab
Description: Tear osmolarity measures the number of milliosmoles of the solutes (e.g., salt) per liter (mOsm/L) of tear. Normal values range from 275 to 295 mOsm/L. Higher values indicate higher concentrations of electrolytes in the tear, which reflect worse dry eye conditions. A diagnosis of dry eye syndrome is made if the osmolarity of either eye is larger than 308 mOsm/L, or when the difference in measured osmolarity between eyes is >8 mOsmol/L
Time Frame: as for outcome 6
Population: All participants receiving both interventions were included in the analysis.
Measure: Mean (Standard Error); unit: mOsm/L (milliosmoles per liter)
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
mOsm/L (milliosmoles per liter) | 302.789 (1.257) | 303.043 (1.257)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Test type: Superiority; p = 0.885, Mixed Models Analysis

10. Secondary Outcome: Dry Eye Measurements (3): Rating of the Corneal Integrity With Lissamine Green Staining (0-4, Lower is Better)
Description: A score on a scale (0-4, lower number indicating a better, healthier cornea); A subjective grade on the Corneal Integrity Rating with Lissamine Green Evaluation Form, which is a clinical grading system used to assess the health and integrity of the corneal surface, particularly focusing on ocular surface damage, dryness, or irritation. It has 5 levels (0-4), with lower numbers being better. Here is the description of each level:
  0: No staining; corneal surface completely intact, no signs of damage. Best possible score.
  1. Minimal staining; few scattered dots of stain, very mild damage or dryness.
  2. Moderate staining; more noticeable punctate staining but no confluent areas.
  3. Marked staining; numerous punctate stains, possible small areas of confluent staining.
  4. Severe staining; large confluent areas of stain, significant epithelial damage. Worst score.
Time Frame: as for outcome 6
Population: All participants receiving both interventions were included in the analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
score on a scale | 2.633 (0.121) | 3.025 (0.125)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Test type: Superiority; p = 0.001, Mixed Models Analysis

11. Secondary Outcome: Dry Eye Measurements (4): Blink Duration (Milliseconds) Measured Through Real-time Blink-contingent Visual Acuity Task
Description: While the subject detected the orientation of a tumbling E, we measured the average interval between two blinks. Larger numbers mean a longer duration of a blink sustained.
Time Frame: as for outcome 6
Population: All participants receiving both interventions were included in the analysis.
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Gunnar OTC Glasses | Control
Number analyzed (Participants) | 35 | 35
milliseconds | 3536.468 (222.0143) | 3514.788 (222.0143)
Statistical Analysis 1: Comparison: Gunnar OTC Glasses vs Control; Test type: Superiority; p = 0.359, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Each subject visited the lab three times: for about 30-40 minutes on visit 1 and about 4 hours each on visits 2 and 3. The adverse events were monitored while the subject was participating in the study for up to 16 days.
Description: Throughout the study, we monitored for adverse events. Minor visual or body discomfort was common for sustained near-distance digital-viewing work and can be relieved by a brief break from the task. So, periodic breaks were put between tasks. Should unusual discomfort not be relieved by a brief break, we would report to the IRB office within 24 hours and give proper modification. No severe or unusual adverse event occurred.
Arm/Group | Gunnar OTC Glasses | Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No